CLINICAL TRIAL: NCT06040190
Title: Evaluation of the Effect of Different Treatments on Pain Scores and Self-reported Oral Health-related Quality of Life in Individuals With Burning Mouth Syndrome: a Randomized Controlled Clinical Trial
Brief Title: Effect of Treatments on Pain and Quality of Life in Individual With Burning Mouth Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Fernando O Costa, Titular Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6.161.933
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Florisil; Clonazepam; Thioctic Acid; Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- topical placebo tablet (Placebo Comparator): magnesium silicate placebo tablet three times a day for 21 days
  Interventions: Drug: topical placebo tablet
- control (No Intervention): artificial saliva
- topical clonazepam tablet (Experimental): 2.0 mg Clonazepam tablet three times a day for 21 days
  Interventions: Drug: topical clonazepam tablet
- oral alpha-lipoic acid capsule (Experimental): 300 mg alpha-lipoic acid capsule twice a day for 60 days
  Interventions: Dietary Supplement: oral alpha-lipoic acid capsule
- topical phytotherapic capsaicin gel (Experimental): 0.025 mg capsaicin gel 4 times a day for 14 days
  Interventions: Other: topical phytotherapic capsaicin gel
- local photobiomodulation (Experimental): Photobiomodulation with wavelength of 810 nm, power of 0.6 W, power density of 1.2 W/cm², beam area of 0.5 cm², and energy of 6 J.
  Interventions: Radiation: local photobiomodulation

INTERVENTIONS:
Drug: topical placebo tablet — Individuals will be instructed to dissolve half a tablet of placebo medication and hold the saliva near the painful oral sites without swallowing, for 3 minutes and then spit. Tablets will contain magnesium silicate, with the same color and flavor as the test medications. Researchers will provide a total of 32 tablets for each participant.
  Other Names: magnesium silicate
  Arms: topical placebo tablet
Drug: topical clonazepam tablet — Individuals will be instructed to dissolve half a tablet of clonazepam and hold the saliva near the painful oral sites without swallowing for 3 minutes and then spit. Researchers will provide a total of 32 tablets for each participant.
  Arms: topical clonazepam tablet
Dietary Supplement: oral alpha-lipoic acid capsule — Participants in this group will be instructed to take oral capsules containing alpha-lipoic acid.
  Arms: oral alpha-lipoic acid capsule
Other: topical phytotherapic capsaicin gel — Participants in this group will to apply the gel containing tocapsaicin on painful oral sites.
  Arms: topical phytotherapic capsaicin gel
Radiation: local photobiomodulation — Photobiomodulation will be applied during 10 seconds per point at 56 points (three on the vestibular mucosa of the 4 quadrants, four on each labial mucosa, six on each of the two buccal mucosae, six on the hard palate, four on each lateral edge of the tongue, six on the dorsum of the tongue, and four sublingual points) with an intermediate distance of 2 mm. A dose of 12 J/cm² per session will be applied in continuous mode for 10 sessions. The 10 sessions will be applied twice a week for 5 consecutive weeks. The LASER will be applied perpendicularly in contact with the mucosa. All patients and the clinician will wear protective glasses.
  Other Names: photodynamic therapy
  Arms: local photobiomodulation

SUMMARY:
Burning Mouth Syndrome (BMS) is characterized by a burning sensation on the tongue or other areas of the mouth, often bilateral but occasionally unilateral. It is more prevalent in postmenopausal women. No specific ethnic or socioeconomic predisposition has been identified. The etiology and pathophysiology of BMS remain unknown. Various treatment approaches have been proposed, yielding conflicting outcomes and underscoring the need for further investigation.

Patients with BMS appear to respond well to long-term therapy involving systemic antidepressants and anxiolytics. The most promising therapeutic effects have been observed with clonazepam, which leads to a significant reduction in pain when applied topically or systemically. Capsaicin, an herbal remedy, also presents as an alternative treatment option, showing positive results in alleviating BMS symptoms when compared to a placebo. Photobiomodulation represents another non-pharmacological treatment possibility. It's analgesic action is possibly attributed to the inhibition of pain mediators. Alpha-lipoic acid (ALA) is dietary supplement employed in BMS treatment. It serves as a potent antioxidant naturally produced within the body, contributing to the mitigation of skin aging and reinforcing the effects of other biological antioxidants. Based on these findings, attempts have been made to demonstrate ALA's effectiveness in BMS management, concluding that ALA may offer benefits in this context.

Therefore, the objective of this study is to investigate, in adults with BMS, the impact of different therapeutic approaches on frequency, intensity, and location of pain, as well as on on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* burning mouth syndrome;
* oral pain that recurs daily for > 2 hours per day for > 3 months;
* pain with burning quality and felt superficially in the oral mucosa;
* oral mucosa appears normal
* oral clinical examination, including sensory tests, is normal;

Exclusion Criteria:

* pregnancy;
* oral mucosal lesions;
* systemic diseases such as diabetes, anemia, deficiency of vitamin B1, B2, B6, B12, Fe, Zinc, and folic acid;
* gastroesophageal reflux;
* previous head and neck radiotherapy;
* Sjogren's disease;
* allergies;
* candidiasis;
* unstimulated saliva flow < 0.25 ml/min and stimulated flow < 1.0 ml/min will be excluded;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | baseline and 3 weeks
  Change in pain scores measured by a visual analog scale and the short version of the McGill Pain Questionnaire. Visual Analogue Scale: values ranging from 0 (no pain) to 10 (most severe pain). The McGill instrument contains 15 descriptors of pain sensation (11 sensory and 4 affective), with each descriptor ranked on a 4-point rating scale (0 = none, 1 = mild, 2 = moderate and 3 = severe). Three measures of pain experience based on sensory and affective descriptors can be obtained: (1) The total index consists of the sum of all 15 descriptors with the total score ranging from 0 to 45; (2) The sensory index consists of the sum of descriptors 1 - 11 with the total score ranging from 0 to 33; and (3) the affective index consists of the sum of descriptors 12 - 15 with the total score ranging from 0 to 12.
Change in pain scores | baseline and 2 months
  Change in pain scores measured by a visual analog scale and the short version of the McGill Pain Questionnaire. Visual Analogue Scale: values ranging from 0 (no pain) to 10 (most severe pain). The McGill instrument contains 15 descriptors of pain sensation (11 sensory and 4 affective), with each descriptor ranked on a 4-point rating scale (0 = none, 1 = mild, 2 = moderate and 3 = severe). Three measures of pain experience based on sensory and affective descriptors can be obtained: (1) The total index consists of the sum of all 15 descriptors with the total score ranging from 0 to 45; (2) The sensory index consists of the sum of descriptors 1 - 11 with the total score ranging from 0 to 33; and (3) the affective index consists of the sum of descriptors 12 - 15 with the total score ranging from 0 to 12.

SECONDARY OUTCOMES:
Change in quality of life scores | baseline and 3 weeks
  Change in quality of life measured by Oral Impacts on Daily Performance scores. Total score ranging from 0 to 275 being classified as: 0 = no impact, values 1 to 10 = low impact, values 11 to 40 = medium impact and values 41 to 275 = high impact (i.e, worse quality of life).
Change in quality of life scores | baseline and 2 months
  Change in quality of life measured by Oral Impacts on Daily Performance scores. Total score ranging from 0 to 275 being classified as: 0 = no impact, values 1 to 10 = low impact, values 11 to 40 = medium impact and values 41 to 275 = high impact (i.e, worse quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando O Costa, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal university of minas gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared.